CLINICAL TRIAL: NCT03034512
Title: Natural History Study of Alpers Huttenlocher Syndrome
Brief Title: Alpers Huttenlocher Natural History Study
Acronym: Alpers
Status: Terminated | Type: Observational
Why Stopped: Research focus has changed.
Sponsor: Columbia University (Other)
Collaborators: Seattle Children's Hospital (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Michio Hirano, MD, Professor of Neurology, Columbia University
Other Study IDs: AAAM9859; 2U54NS078059-04 (NIH); 5U54NS078059-02 (NIH)
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Alpers Huttenlocher Syndrome
MeSH Terms: conditions — Diffuse Cerebral Sclerosis of Schilder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Alpers-Huttenlocher: Patients confirmed to have Alpers Huttenlocher Syndrome
- Siblings: Siblings of patients with Alpers Huttenlocher Syndrome

SUMMARY:
This is a natural history study of Alpers Huttenlocher Syndrome. Patients will be followed over time to assess clinical symptoms for the purpose of expanding knowledge of this disorder in the medical community.

DETAILED DESCRIPTION:
The study team will conduct outpatient visits to the medical center on a 6 month basis, or as patients are able. The patients or their caregivers will complete medical and symptom questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* All individuals of any age with confirmed Alpers Huttenlocher Syndrome (AHS) or siblings of confirmed AHS patients are eligible to participate. AHS requires the presence of polymerase gamma 1 (POLG) pathological mutations, either homozygous or compound heterozygote mutations, and the presence of epilepsy and either, developmental regression or hepatopathy. If POLG mutations are not demonstrated, AHS requires the presence of refractory seizures, developmental regression, and hepatopathy as well as two or more other clinical and laboratory findings including elevated cerebrospinal fluid (CSF) protein, neuroimaging showing lactate peaks, reduced N-acetyl aspartate with hyperintensities on T2/FLAIR in the thalamus and posterior head regions, optic atrophy/cortical blindness, quantitative mtDNA reduction (>30% ) in muscle and/or liver, non-specific electron transport chain (ETC) enzyme deficiencies.
* All patients must agree to participate in the North American Mitochondrial Disease Consortium (NAMDC) Clinical Registry

Exclusion Criteria:

* Patient does not have confirmed AHS and is not the sibling of a patient with confirmed AHS
* Not willing to participate in the NAMDC clinical Registry

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients with Alpers Huttenlocher Syndrome (AHS) and their siblings
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
onset age | 2 years
  age at onset of first symptom versus POLG mutation type

CONTACTS AND LOCATIONS:
Overall Officials: Michio Hirano, MD, Principal Investigator — Columbia University; Russell Saneto, MD, Study Chair — Seattle Children's Hospital
Locations (2):
- United States (2):
  - Columbia University, New York, New York
  - Seattle Childrens Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
This study is a sub project under the North American Mitochondrial Disease Consortium. The de-identified data can be shared if investigators have Institutional Review Board (IRB) approval for a project that might include data from this study and if the NAMDC administration approves of the project

REFERENCES:
- See also: North American Mitochondrial Disease Consortium (NAMDC) Study Site — https://www.rarediseasesnetwork.org/cms/namdc/Get-Involved/Studies/7405